CLINICAL TRIAL: NCT03932097
Title: Feasibility of a Mobile Parent-based Intervention to Reduce Alcohol Use by High School Seniors
Brief Title: REAL Parenting Alcohol and Substance Use App
Acronym: RP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Prevention, LLC (Industry)
Responsible Party: Principal Investigator, Michael Hecht, President, Real Prevention, LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11690
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Underage Drinking; Alcohol Use, Underage
MeSH Terms: conditions — Underage Drinking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL Parenting (Experimental): REAL Parenting digital intervention emphasizing parent-teen/young adult communication on drinking/risks of drinking/risks of alcohol abuse, with the addition of a communication component on the risks of nicotine and marijuana use, with the goal of reducing alcohol, nicotine and marijuana use in college students.
  Interventions: Behavioral: REAL Parenting
- Active Control Materials (Active Comparator): NIAAA materials on underage drinking for parents
  Interventions: Other: Active Control Materials

INTERVENTIONS:
Behavioral: REAL Parenting — REAL Parenting digital intervention emphasizing parent-teen/young adult communication on drinking/risks of drinking/risks of alcohol abuse, with the addition of a communication component on the risks of nicotine and marijuana use, with the goal of reducing alcohol, nicotine and marijuana use in college students.
  Arms: REAL Parenting
Other: Active Control Materials — NIAAA materials on underage drinking for parents
  Arms: Active Control Materials

SUMMARY:
High school students' alcohol, nicotine, and marijuana use are major public health problems. Among the many consequences of these risky behaviors are impaired driving and impaired passenger fatalities as well as increased health risks. Both school administrators and parents have requested parent-based interventions (PBIs)for the general high school population that include content on alcohol, nicotine and marijuana use. In addition, digital materials are needed for the "on-the-go" parent. The proposed research will address this omission, curb the alarming trends noted above, and move the field forward by conducting a randomized controlled trial testing a modified, digital version of the Parent Handbook for the all high school students that includes additional content for parents to have broader discussions about combined alcohol nicotine and marijuana use alone (referred to as REAL Parenting). Parent-teen dyads will be invited to participate and complete baseline assessment and parents will receive the REAL Parenting or active control materials shortly afterwards. This will allow an examination of the impact of the RP on alcohol use, and associated consequences and sustained effects across the follow-up period.

DETAILED DESCRIPTION:
The goal of this Phase II SBIR is to provide an efficient, engaging, and effective means to enhance parents' ability to reduce prevalence of alcohol use and consequences, and other substance use through the development and evaluation of REAL Parenting (RP). RP is a brief, interactive, self-paced, and digital curriculum for parents of high-school-aged adolescents, a frequently neglected population created from the evidence-based Parent Handbook,available in hard copy and DVD for college-bound youth only. The curriculum is needed because most parent-based prevention interventions target children or young adolescents, neglecting older adolescents, despite that fact that alcohol use increases in frequency and risk through midadolescence. Also, unlike other evidence-based parenting curricula, RP is brief, requires only the parents, does not require training, and can be used "on the go" through any digital device. This provides a market niche for the proposed project that addresses this curriculum gap through the innovative use of both technology and prevention science. This format will allow us to personalize or target parents based on their communication style and allows parents to customize their experience by choosing or clicking through the optional content. Personalization and customization are two essential engagement strategies for digital prevention interventions.

ELIGIBILITY:
Inclusion Criteria:

* High school students (ages 15-18) who may be at risk for alcohol, marijuana and nicotine use and abuse, and whose parent/guardian is willing to participate in the proposed study as part of a parent/student dyad.
* High school students ages 15-18 with their parents/guardians; English fluency; Internet access; at least one parent/guardian fluent in English and with Internet access

Exclusion Criteria:

* Not high school aged (not ages 15-18)
* Parent/guardian was not willing to participate
* Does not have English fluency;
* Does not have access to Internet access

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 306 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | Project years 1-2
  A standard drink definition will be provided: a standard drink consists of 12 oz. beer or wine cooler, 8.5 oz. of malt liquor, 4 oz. of wine, 3.5 oz. fortified wine, or 1.5 oz. of hard liquor. Typical weekly drinking: participants will respond to the Daily Drinking Questionnaire(DDQ; Collins et al., 1985) to indicate number of drinks consumed on each day of a typical week within the past six months. Participants will report maximum number of drinks consumed on an occasion within the past month and number of hours spent drinking on that occasion using the Quantity/Frequency/Peak questionnaire (QFP; Dimeff et al., 1999; Marlatt et al., 1998). Drunkenness will be assessed by asking how many times in the past month participants have gotten drunk, or very high from alcohol using a 6-point scale: (0) never to (5) 9 or more. Heavy episodic drinking will be measured for females and males separately, asking for number of times they?ve had 4/5, respectively, drinks in a row within two hours.

SECONDARY OUTCOMES:
Marijuana Use | Project years 1-2
  Frequency of use will be assessed by asking how often participants used marijuana during the past six months using a 7-point scale ranging from (0) never to (6) 40 or more times.
Combined Use | Project years 1-2
  Frequency of combined use will be assessed for participants indicating marijuana and nicotine use with a single item: During times you used marijuana, how often did you also drink alcohol? using a 6-point scale ranging from (0) never to (5) 40 or more times. For participants that indicate their peak drinking occasion a follow up question will assess whether marijuana or nicotine was also used(yes or no).
Consequences of Alcohol Use | Project years 1-2
  Alcohol-related consequences (e.g., said or done embarrassing things, blackout) from the past six months will be measured using the established Brief Young Adult Alcohol Consequences Questionnaire (BYAACQ; Read, Kahler, Strong, & Colder, 2006). Response options will again be measured on the same a 7-point scale as Combined Use.
Nicotine Use | Project years 1-2
  Frequency of use will be assessed by asking how often participants used nicotine products (tobacco, vaping, snuff) during the past six months using a 7-point scale ranging from (0) never to (6) 40 or more times.

OTHER OUTCOMES:
Alcohol Motives | Project years 1-2
  Using the past six months as a time reference, participants will be asked about their motivations to use alcohol. Twenty items for each substance will assess motives for using alcohol, such as "to be sociable" and "to forget about your problems" on a 5-point scale ranging from (1) almost never/never to (5) almost always/always.
Alcohol Expectancies | Project years 1-2
  Alcohol expectancies will be measured using a 7-point scale ranging from (-3) strongly disagree to (3) strongly agree. Items will assess how likely a variety of alcohol-related consequences will be experienced in the next few months. For example, items, be worded specifically for alcohol use, such as "I will feel badly about myself because of my drinking."
Alcohol Willingness | Project years 1-2
  Response options for willingness items will be on a 7-point scale ranging from (1) strongly disagree to (7) strongly agree. Willingness to use alcohol will be measured to assess participants? willingness to 1) drink once or twice in two hours; 2) drink 3-4 times in two hours; and 3) drink 5+ times in two hours. Willingness to use marijuana and COMBINE will be assessed individually with four items asking their willingness to use marijuana/COMBINE occasionally, regularly, weekly, and daily.
Alcohol Norms | Project years 1-2
  Perceived norms of drinking for the past six months will be measured using the DDQ using closest friend as a referent. To assess peer injunctive norms of alcohol use participants will be asked to indicate how acceptable their closest friends would find of a list of situations (e.g., drinking enough alcohol to pass out) using a (1) strongly disapprove to (7) strongly approve scale.
Parental Communication | Project years 1-2
  Parental communication about alcohol, nicotine, and marijuana use, COMBINE, and alcohol consequences will be assessed separately for parent and teen. Participants will be asked whether their parent discussed these topics (yes/no) with them within the past six months. Items include topics such as "the importance of not being pressured to drink to fit in" and "how marijuana works in the body."

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hecht, Principal Investigator — REAL Prevention
Locations (1):
- REAL Prevention, LLC, Clifton, New Jersey, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/97/NCT03932097/Prot_SAP_000.pdf